CLINICAL TRIAL: NCT02956356
Title: Acute Effects of SATIOSTAT Ingestion on Satiation Hormones, Gastric Emptying, Subjective Feelings of Appetite and Energy Intake
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: SATIOSTAT acute effects
Record Dates: First submitted 2016-11-02; First posted 2016-11-07 (Estimated); Last update posted 2018-08-08 (Actual); Status verified 2018-08

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — Glucose; CD36 Antigens; Carbohydrates; Proteins

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- Control treatment + oral glucose (Placebo Comparator): Control treatment as preload and then an oral glucose load of 75g enriched with C13 sodium acetate (for determination of gastric emptying rates)
  Interventions: Dietary Supplement: Control treatment + oral glucose
- SATIOSTAT treatment + oral glucose (Active Comparator): SATIOSTAT treatment as preload and then an oral glucose load of 75g enriched with C13 sodium acetate (for determination of gastric emptying rates)
  Interventions: Dietary Supplement: SATIOSTAT treatment + oral glucose
- Control treatment + meal intake (Placebo Comparator): Control treatment as preload followed by a test meal
  Interventions: Dietary Supplement: Control treatment + meal intake
- SATIOSTAT treatment + meal intake (Active Comparator): SATIOSTAT treatment as preload followed by a test meal
  Interventions: Dietary Supplement: SATIOSTAT treatment + meal intake

INTERVENTIONS:
Dietary Supplement: Control treatment + oral glucose — Control granulates (maize starch and long-chain fatty acids) with powder; 75g oral glucose load
  Other Names: The energy content of one single bottle control is 138kcal and contains 7.6g fat, 11.1g carbohydrates and 3.9g protein.
  Arms: Control treatment + oral glucose
Dietary Supplement: SATIOSTAT treatment + oral glucose — SATIOSTAT granulates (hydrocolloids (fibers) and long-chain fatty acids) with powder; 75g oral glucose load
  Other Names: The energy content of one single bottle SATIOSTAT is 138kcal and contains 10.5g fat, 6.4g carbohydrates and 3.9g protein.
  Arms: SATIOSTAT treatment + oral glucose
Dietary Supplement: Control treatment + meal intake — Control granulates (maize starch and long-chain fatty acids) with powder; test meal (ham sandwiches: 50g bread, 10g butter, 29g ham (pork); 247 kcal/sandwich) and tap water)
  Other Names: The energy content of one single bottle control is 138kcal and contains 7.6g fat, 11.1g carbohydrates and 3.9g protein.
  Arms: Control treatment + meal intake
Dietary Supplement: SATIOSTAT treatment + meal intake — SATIOSTAT granulates (hydrocolloids (fibers) and long-chain fatty acids) with powder; test meal (ham sandwiches: 50g bread, 10g butter, 29g ham (pork); 247 kcal/sandwich) and tap water)
  Other Names: The energy content of one single bottle SATIOSTAT is 138kcal and contains 10.5g fat, 6.4g carbohydrates and 3.9g protein.
  Arms: SATIOSTAT treatment + meal intake

SUMMARY:
SATIOSTAT is a composition comprising a specific dietary fibre component (a mixture of hydrocolloids with excellent safety profiles and a long history of use in humans) and a lipid component (long-chain fatty acids). The goal of this combination is to achieve long-acting delivery of long-chain fatty acids to the intestinal lining, triggering the sustained release of satiety-signals from intestinal cells, and consequently reducing appetite and lowering food intake in humans.

Effects of acute ingestion of SATIOSTAT vs. a control will be examined. On a first and second study day, volunteers receive a preload of either SATIOSTAT or a control and then an oral glucose load of 75g enriched with C13 sodium acetate. Gastric emptying will be measured by means of a breath test, and insulin, glucose and satiation hormones will be assessed. On the third and fourth study day, volunteers receive a preload of either SATIOSTAT or a control and are then presented a test meal. Total calorie intake is measured as well as subjective feelings of satiation. In addition satiation hormones are measured.

ELIGIBILITY:
Inclusion Criteria:

* Obese volunteers (BMI > 30kg/m2)
* Otherwise healthy
* Informed Consent as documented by signature (Appendix Informed Consent Form)

Exclusion Criteria:

* Food allergies, food intolerance
* Evidence of relevant cardiovascular, pulmonary, renal, hepatic, pancreatic, gastrointestinal, metabolic, endocrinological, neurological, psychiatric or other diseases at screening
* Chronic or clinically relevant acute infections
* Clinically relevant abnormalities in chemical, haematological or any other laboratory parameters
* Participation in drug trials within 2 months before start of the study
* Neurological or psychiatric disease or drug or alcohol abuse, which would interfere with the subjects proper completion of the protocol assignment
* Pregnancy: although no contraindication pregnancy might influence metabolic state. Women who are pregnant or have the intention to become pregnant during the course of the study are excluded. In female participants of childbearing age not using safe contraception (oral, injectable, or implantable contraceptives, or intrauterine contraceptive devices) a urine pregnancy test is carried out upon screening.
* Antibiotic therapy within the last 3 months before inclusion
* Substance abuse, alcohol abuse
* Inability to follow procedures due to psychological disorders, dementia or insufficient
* Knowledge of project language (German).
* Participation in another study with investigational drug within the 30 days preceding and during the present study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2016-10; Primary Completion 2018-02 (Actual); Study Completion 2018-02 (Actual)

PRIMARY OUTCOMES:
Acute effects of SATIOSTAT on gastrointestinal (GI) peptide release measured by ELISA | changes from baseline to three hours after treatment
  measured by commercially available ELISA (enzyme-linked immunosorbent assay )-kits

SECONDARY OUTCOMES:
Acute effects of SATIOSTAT on glucose tolerance measured by oral glucose tolerance test | changes from baseline to three hours after treatment
  measured with oral glucose tolerance test
Acute effects of SATIOSTAT on gastric emptying measured by 13C-sodium-acetate breath test | changes from baseline to four hours after treatment
  measured by 13C-sodium-acetate breath test
Acute effects of SATIOSTAT on subjective feelings of hunger and satiety measured by visual analogue scales | changes from baseline to three hours after treatment
  measured by visual analogue scales
Acute effects of SATIOSTAT on subsequent calorie intake measured by calorie intake from a test meal | changes from baseline to two hours after treatment
  calorie intake from a test meal will be assessed

CONTACTS AND LOCATIONS:
Overall Officials: Christoph Beglinger, MD, Study Chair — St. Claraspital klinische Forschungsabteilung
Locations (1):
- St Claraspital, Basel, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided